CLINICAL TRIAL: NCT06539832
Title: Correlation Analysis of Intestinal Flora and Immune Function in Patients With Monoclonal Immunoglobulinaemia Co-infection
Brief Title: Intestinal Flora and Immunity in Monoclonal Gammopathy Patients
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZhujiangMGUS
Record Dates: First submitted 2024-07-22; First posted 2024-08-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma; MGUS; Gut Microbiota; Infections; M-Protein
MeSH Terms: conditions — Multiple Myeloma; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Monoclonal gammopathy patients without concurrent infection: (I) Inclusion criteria:
  1. Age 45 years or older;
  2. Patients screened positive for monoclonal protein by MALDI-TOF MS;
  3. No symptoms of infection, with normal infection indicators (whole blood hs-CRP, serum IL-6, PCT);
  4. Adequate remaining whole blood, plasma and stool samples available, and relevant case data can be provided.
  (II) Exclusion criteria:
  1. History of intestinal tumors, irritable bowel syndrome or inflammatory bowel disease, or diagnosed during hospitalization;
  2. Received antibiotic treatment in the past one month;
  3. Insufficient sample volume, or presence of severe hemolysis, lipemia, jaundice or other unqualified sample conditions.
- Monoclonal gammopathy patients with concurrent infection: (I) Inclusion criteria:
  1. Age 45 years or older;
  2. Patients screened positive for monoclonal protein by MALDI-TOF MS;
  3. Presence of infection symptoms, with abnormal infection indicators (whole blood hs-CRP, serum IL-6, PCT);
  4. Adequate remaining whole blood, plasma and stool samples available, and relevant case data can be provided.
  (II) Exclusion criteria:
  1. History of intestinal tumors, irritable bowel syndrome or inflammatory bowel disease, or diagnosed during hospitalization;
  2. Received antibiotic treatment in the past one month;
  3. Insufficient sample volume, or presence of severe hemolysis, lipemia, jaundice or other unqualified sample conditions.
- Healthy control group: (I) Inclusion criteria:
  1. Age 45 years or older;
  2. Patients screened negative for monoclonal protein by MALDI-TOF MS;
  3. No symptoms of infection, with normal infection indicators (whole blood hs-CRP, serum IL-6, PCT);
  4. Adequate remaining whole blood, plasma and stool samples available, and relevant case data can be provided.
  (II) Exclusion criteria:
  1. History of intestinal tumors, irritable bowel syndrome or inflammatory bowel disease, or diagnosed during hospitalization;
  2. Received antibiotic treatment in the past one month;
  3. Severe systemic diseases including malignant tumors;
  4. Insufficient sample volume, or presence of severe hemolysis, lipemia, jaundice or other unqualified sample conditions.

SUMMARY:
This study aims to investigate the characteristics of the gut microbiota and immune function status in patients with monoclonal gammopathy complicated by infection, and to analyze the correlation between the two.200 patients diagnosed with monoclonal gammopathy by MALDI-TOF MS were included, of which 100 had concurrent infections and 100 did not. An additional 100 healthy controls, matched for age and gender, were also enrolled.By comparing the composition of the gut microbiota and immune function markers (such as peripheral blood immune cell profiles and cytokine levels) between the patient groups and the control group, the study will evaluate the dysbiosis of the gut microbiota and abnormal immune status in patients with monoclonal gammopathy complicated by infection. The aim is to explore the correlation between the gut microbiome alterations and immune dysfunction, in order to provide a basis for further investigation of the underlying mechanisms.

DETAILED DESCRIPTION:
The intestine is the largest immune organ in the human body, playing a crucial role in regulating host health, maintaining metabolic and immune homeostasis, and preventing pathogen invasion. The gut microbiota can directly participate in the immune regulation of the host, promote the development of the immune system, and maintain normal immune function. Meanwhile, the immune system also has a regulatory and constraining effect on the gut microbiota. With age, the structure of the gut microbiota and the function of the immune system undergo continuous changes and adjustments to adapt to the body's needs. This dynamic gut microbiota-immune system interaction plays a key role in maintaining metabolic homeostasis and immune balance in the body.Multiple myeloma (MM) is a hematological malignancy characterized by the clonal proliferation of malignant plasma cells in the bone marrow, commonly seen in middle-aged and elderly individuals. MM patients generally have a higher risk of infection, especially after receiving intensive chemotherapy or hematopoietic stem cell transplantation.Monoclonal gammopathy of undetermined significance (MGUS) is an asymptomatic condition, and multiple myeloma often progresses from monoclonal gammopathy. Although most MGUS patients do not progress to malignant disease for life, MGUS patients do have a higher risk of infection. Gut microbiome dysbiosis may be involved in regulating immune function, leading to increased susceptibility to infections in MGUS patients.This study aims to use a retrospective cohort study approach to systematically analyze the characteristics of the gut microbiota in MGUS patients with concurrent infections, and explore its correlation with immune-related indicators. In-depth analysis of these key factors will help further elucidate the pathogenesis of MGUS complicated by infection, and provide new evidence and insights for clinical prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 years and older; and
2. Patients who were monoclonal gammaglobulin negative by MALDI-TOF MS screening;
3. No symptoms of infection and normal indicators of infection (whole blood hs-CRP, serum IL-6, PCT);
4. Sufficient remaining whole blood, plasma and faecal samples are available, and relevant case information can be provided.

Exclusion Criteria:

1. Those with a previous history of intestinal tumour, irritable bowel syndrome or inflammatory bowel disease or confirmed in hospital; and
2. Patients receiving antibiotic therapy in the last month
3. Severe systemic diseases including malignant tumours;
4. Insufficient remaining sample volume, or the presence of sample failure such as severe haemolysis, lipaemia or jaundice.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients aged 45 years and older who meet the following inclusion criteria:
  1. Monoclonal gammopathy negative as determined by MALDI-TOF MS screening.
  2. No symptoms of infection and normal levels of inflammatory markers (whole blood hs-CRP, serum IL-6, PCT).
  3. Availability of sufficient remaining whole blood, plasma and fecal samples, as well as relevant case information.
  Patients will be excluded if they have:
  1. A previous history of intestinal tumors, irritable bowel syndrome or inflammatory bowel disease.
  2. Received antibiotic therapy within the last month.
  3. Severe systemic diseases, including malignant tumors. Insufficient sample volume or presence of sample failure (e.g. severe hemolysis, lipemia or jaundice).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
M-protein detection | 24 months
  Plasma samples from all patients will be screened and qualitatively analysed for M proteins using MALDI-TOF MS to determine the presence of patients with monoclonal gammaglobulinemia.
microbiome | 24 months
  To assess the value of the microbiome in predicting the prognosis of patients with monoclonal gammopathy and in diagnosing co-morbidities. To analyse the microbial composition of patient stool samples using 16S rRNA gene sequencing and metagenomics.
immunological function | 24 months
  To assess the number and function of peripheral blood immune cells (T-cells, B-cells, NK-cells, etc.) in patients with monoclonal gammaglobulinaemia. To further investigate the potential therapeutic value of intestinal microecological modulation in improving the immune status of MGUS patients.
metabonomics | 24 months
  To assess changes in plasma metabolomics in patients with monoclonal gammaglobulinaemia. Metabolomics is a large-scale study of small molecules such as fatty acids, bile acids, and lipid mediators.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, Professor, Study Chair — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No